CLINICAL TRIAL: NCT02628977
Title: Tailored Peer-Based Sleep Health Education and Social Support Among Blacks With Obstructive Sleep Apnea
Brief Title: Sleep Health Education and Social Support Among Blacks With OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-01028; NCT02427815 (obsolete NCT alias)
Record Dates: First submitted 2015-12-08; First posted 2015-12-11 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OSA Health Education & Support Group (Experimental): Participants randomly assigned to the intervention arm will receive OSA health education and social support from a trained Peer educator.
  Interventions: Behavioral: Peer Based Sleep Health Education and Social Support
- Attention Control Group (Active Comparator): Participants in the attention control group will receive standard sleep literature, providing information about Obstructive Sleep Apnea and access to available sleep services.
  Interventions: Behavioral: Attention Control Group

INTERVENTIONS:
Behavioral: Peer Based Sleep Health Education and Social Support — Participants randomly assigned to the intervention arm will receive Obstructive Sleep Apnea education and social support from a trained Peer Educator.
  Arms: OSA Health Education & Support Group
Behavioral: Attention Control Group — Participants assigned to this arm of the study will receive standard sleep literature, providing information about OSA and access to available sleep services.
  Arms: Attention Control Group

SUMMARY:
The primary purpose of this study is to ascertain the effectiveness of tailored, peer based sleep health education and social support in increasing adherence rates to recommended Obstructive Sleep Apnea (OSA) evaluation and treatment among blacks at risk of Obstructive Sleep Apnea.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA), which disproportionately affects blacks (31% vs. 10%, whites), is a critical, preventable and/or treatable disease potentially causing increased cardiovascular disease (CVD) outcomes (e.g., obesity, diabetes, hypertension, stroke, arrhythmia, and chronic heart failure). Improving sleep may have direct effects in reducing CVD risk,2 enhancing brain functions, and increasing workplace productivity. Unfortunately, our focus groups suggest that most at-risk blacks are unaware of OSA symptoms or its related morbidity. Thus, it is imperative to address poor adherence among blacks with OSA, if we are to reduce health disparities associated with CVD outcomes between blacks and whites.

This is a randomized study with a total of 6 sites recruiting; 3 will serve as controls and 3 that will be intervention. Group A participants (Intervention group) will receive health education from a trained Peer Health Educator and Group B participants (Control group) will meet with a salon worker, barbershop worker, or church Health Ministry group leader. Participants will be asked to use a sleep diary and wear a home sleep test device to measure sleep for 7 days. They will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* self-reported race/ethnic minority
* ages ≥18 years
* accessible by telephone
* consent to participate, which includes permission to release medical record information
* A positive screening for OSA is necessary to be enrolled in the intervention protocol.

Exclusion Criteria:

* are involved in another sleep study.
* are unable to understand and sign this informed consent form.
* know someone who is participating in this study.
* had a heart attack or stroke within the past 12 weeks.
* do not identify yourself as a racial/ethnic minority.
* are pregnant.
* Refuse to use the ARESTM home sleep test device.
* Refuse to use the WatchPATTM home sleep test device.
* are not at risk for sleep apnea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1092 (Actual)
Dates: Start 2015-11; Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Rate of adherence to recommended home OSA evaluation and treatment after intervention exposure | 12 Months
  We will perform analysis on an intention-to-treat basis.

SECONDARY OUTCOMES:
Rate of Obstructive Sleep Apnea among black men and women at the community level | 12 Months
  Obstructive Sleep Apnea among minorities.

CONTACTS AND LOCATIONS:
Overall Officials: Girardin Jean Louis, MD, Principal Investigator — New York University Medical School
Locations (1):
- 180 Madison Ave, New York, New York, United States

REFERENCES:
- [Derived] Seixas AA, Trinh-Shevrin C, Ravenell J, Ogedegbe G, Zizi F, Jean-Louis G. Culturally tailored, peer-based sleep health education and social support to increase obstructive sleep apnea assessment and treatment adherence among a community sample of blacks: study protocol for a randomized controlled trial. Trials. 2018 Sep 24;19(1):519. doi: 10.1186/s13063-018-2835-9. PMID 30249293